CLINICAL TRIAL: NCT00641199
Title: The Effect of Jarro-Dophilus EPS Probiotics on the Prevention of Diarrhea, Quality of Life and Symptoms in Adults Receiving Antibiotic Therapy.
Brief Title: Probiotics for Prevention of Antibiotic-associated Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Jarrow Formulas Inc (Industry); Institut Rosell (Other)
Responsible Party: Yvonne M. Shevchuk, B.S.P., Pharm D, College of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAAD-07-112; 07-112
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Antibiotic-Associated Diarrhea
Keywords: Antibiotic-associated diarrhea; Probiotic; Quality of life; Antibiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Jarrow-Dophilus EPS
  Interventions: Other: Jarro-Dophilus EPS probiotics
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Jarro-Dophilus EPS probiotics

INTERVENTIONS:
Other: Jarro-Dophilus EPS probiotics — Jarro-Dophilus EPS product 2 capsules twice daily. 4.4 billion live bacteria per capsule.

SUMMARY:
The purpose of this study is to evaluate if ingestion of a probiotic formula (Jarrow-Dophilus EPS)reduces incidence of diarrhea and improves the quality of life of patients receiving antibiotic therapy.

DETAILED DESCRIPTION:
A common complication of antibiotic use is antibiotic-induced diarrhea (AAD). AAD is the result of disrupted microflora, occurring two to eight weeks after antibiotic use. Probiotic supplementation may rebalance the intestinal flora, thus reducing the incidence of diarrhea, improving quality of life and reducing symptoms associated with antibiotic administration.

The proposed study will be a prospective, randomized, double blind, placebo-controlled trial that will assess the efficacy of the Jarro-Dophilus EPS probiotics formula for the prevention of AAD.

In addition,a subgroup of participants will be requested to provide one fecal sample at the initiation of the study and one sample in the last three days of probiotic (or placebo) treatment. The samples will undergo microbial analysis for routine C & S(Salmonella, Shigella, Campylobacter, Ecoli 0157, Yersinia), VRE, Yeast, Fungus culture (moulds) and C. difficile toxin.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Prescribed oral or IV antibiotics by physicians in Saskatoon Health Region's community medical clinics

Exclusion Criteria:

* Treatment with an antibiotic two weeks prior to study entry
* Underlying long term gastrointestinal disease (i.e., Ulcerative Colitis, Crohn's Disease, irritable bowel syndrome, ileostomy, colostomy)
* Pregnant or lactating
* Immunocompromised state
* Chronic illness such as Hepatitis B, Hepatitis C, renal failure
* Inability to provide informed consent, inability to speak or write in English
* Receiving tube feeds
* Insufficiently functional (physically and cognitively) to complete the study diary and questionnaires.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of patients experiencing diarrhea | Duration of antibiotic course plus 3 weeks

SECONDARY OUTCOMES:
Duration of diarrhea | Duration of antibiotic course plus 3 weeks
Quality of life. | Duration of antibiotic course plus 3 weeks
Gastrointestinal Symptom Rating Scale score. | Duration of antibiotic course plus 3 weeks
Incidence of adverse effects. | Duration of antibiotic course plus 3 weeks
Presence of pathogens in fecal samples. | Duration of antibiotic course

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M Shevchuk, B.S.P., Pharm D., Principal Investigator — College of Pharmacy and Nutrition, University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada